CLINICAL TRIAL: NCT05041699
Title: A Randomized, Double-Blind, Phase 1b Study in Healthy HIV-Negative Women to Evaluate the Pharmacokinetics, Safety, and Bleeding Patterns Associated With 90-Day Use of Core-Sheath Vaginal Rings Releasing Dapivirine and Levonorgestrel
Brief Title: PK, Safety Study of 90-Day Use of Vaginal Rings Containing Dapivirine and Levonorgestrel
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: International Partnership for Microbicides, Inc. (Industry)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: IPM 056/CCN019B
Record Dates: First submitted 2021-08-24; First posted 2021-09-13 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-03

CONDITIONS: Pharmacokinetics; Safety Issues; Bleeding
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IPM Ring-105 (Experimental): Ring-105 (xx mg dapivirine + xxx mg levonorgestrel)
  Interventions: Combination Product: IPM Ring-105
- IPM Ring-106. (Active Comparator): Ring-106 (xx mg dapivirine + xxx mg levonorgestrel)
  Interventions: Combination Product: IPM Ring-106

INTERVENTIONS:
Combination Product: IPM Ring-105 — DPV-LNG Ring containing xx mg of dapivirine + xx mg of levonorgestrel
  Arms: IPM Ring-105
Combination Product: IPM Ring-106 — DPV-LNG Ring containing xx mg of dapivirine + xx mg of levonorgestrel
  Arms: IPM Ring-106.

SUMMARY:
A double-blind, randomized trial (1:1) to characterize the local and systemic pharmacokinetics (PK) of two DPV-LNG vaginal ring formulations

DETAILED DESCRIPTION:
A Randomized, Double-Blind, Phase 1b Study in Healthy HIV-Negative Women to Evaluate the Pharmacokinetics, Safety, and Bleeding Patterns Associated with 90-Day Use of Core-Sheath Vaginal Rings Releasing Dapivirine and Levonorgestrel

ELIGIBILITY:
Inclusion Criteria:

1. Assigned female sex at birth Note: Participants who are female at birth, who now identify as male, will not be excluded so long as they are not currently or have not been on female-to-male transition therapy within 90 days prior to Enrollment
2. Age 18 through 45 years (inclusive) at Screening
3. Able and willing to provide written informed consent to be screened for and enrolled in the CCN019B study
4. Able and willing to provide adequate locator/contact information
5. Able to communicate in spoken and written English
6. Available for all visits and able and willing to comply with all study procedures and requirements
7. Willing to abstain from insertion of anything into the vagina (including receptive intercourse, tampons) for 24 hours preceding the Enrollment Visit and clinical visits where samples are taken
8. Not at risk for pregnancy due to use of an effective nonhormonal method of contraception or practice per participant report at Enrollment, and intending to continue use of an effective, non-hormonal method for the duration of study participation. Effective methods and practices are defined as:

   1. Non-hormonal (e.g. copper) intrauterine device (IUD) inserted at least 90 days prior to Enrollment
   2. Consistent and correct male condom use*

      *Details regarding this criterion will be specified in the IPM 056/CCN019B Study Manual
   3. Sterilization (of participant or partner)
   4. Having sex exclusively with individuals assigned female sex at birth
   5. Sexually abstinent for 90 days prior to Enrollment, and intending to remain abstinent for the duration of study participation
   6. Permanent contraception
9. In general, good health as determined by the Investigator of Record (IoR)/designee at Screening and Enrollment visits
10. HIV-uninfected based on testing performed at the Screening and Enrollment visits
11. Per participant report at Screening, current regular menstrual cycles of approximately 21 to 35 days in duration with no reported intermenstrual bleeding or heavy menstrual bleeding per discussion with the Investigator.
12. Intact uterus with at least one ovary
13. Per participant report at Screening and Enrollment visits, states a willingness to refrain from inserting any non-study vaginal products or objects into the vagina from the Enrollment Visit through completion of the in-person PK follow-up visits with the exception of tampon use and intercourse, which can occur but not within 24 hours of the study visit.
14. Documentation of a satisfactory Pap test within ASCCP or ACOG guidelines such that additional treatment will not be required during the study period. If a copy of a Pap test (and indicated follow-up testing) is not available and the subject is 21 years or older, a Pap test should be done during the screening period.
15. Subjects must be ovulatory as confirmed by a documented screening progesterone (P4) level ≥ 3 ng/mL by local laboratory.
16. At Screening and Enrollment visits, agrees not to participate in other research studies involving drugs, medical devices, vaginal products or vaccines after the Screening Visit through completion of participation on the trial.

Exclusion Criteria:

1. BMI greater than 40 kg/m2 at Screening visit
2. Pregnant at Screening or Enrollment visits or plans to become pregnant during the study period Note: A documented negative pregnancy test performed by study staff is required for inclusion; however, a self-reported pregnancy is adequate for exclusion from the study.
3. Diagnosed with symptomatic urinary tract infection (UTI) or reproductive tract infection (RTI) at Screening or Enrollment visits. Otherwise eligible participants diagnosed with symptomatic UTI/RTI during screening will be offered treatment. If treatment is complete and symptoms have resolved within the 90-day screening window, eligible participants may be enrolled.
4. Diagnosed with an acute STI requiring treatment per current CDC guidelines (http://www.cdc.gov/std/treatment/) at Screening or Enrollment visits such as gonorrhea (GC), chlamydia, trichomonas, and/or pelvic inflammatory disease (PID) Note: Genital warts requiring treatment and greater than two disease flares of herpes simplex virus (HSV) within a year are considered exclusionary; however, infrequent HSV outbreaks are not. Genital warts requiring treatment are defined as those that cause undue burden or discomfort to the participant, including bulky size, unacceptable appearance, or physical discomfort. See IPM 056/CCN019B Study Manual for additional information.
5. Has a clinically apparent Grade 2 or higher pelvic exam finding (observed by study staff) at Screening or Enrollment, as per the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017, and/or Addendum 1 (Female Genital Grading Table for Use in Microbicide Studies [Dated November 2007]) Note: Cervical bleeding associated with speculum insertion and/or specimen collection judged to be within the range of normal according to the clinical judgment of the IoR/designee is considered expected non-menstrual bleeding and is not exclusionary.

   Note: Otherwise eligible participants with exclusionary pelvic exam findings may be enrolled/randomized after the findings have improved to a non-exclusionary severity grading or resolved within 90 days of providing informed consent for screening.
6. Participant report and/or clinical evidence of any of the following:

   1. Known adverse reaction to any component of the study product (ever)
   2. Chronic and/or recurrent vaginal candidiasis and/or recurrent symptomatic bacterial vaginosis
   3. Has a contraindication to a progestin-only contraceptive method as defined by a category 3 or 4 condition according to the CDC US Medical Eligibility Criteria for Contraceptive Use, 201652
   4. Use of hormonal contraception, including hormonal IUD and implants within the 28 days prior to the Enrollment Visit.
   5. Current use or planned use of strong CYP3A inhibitors and inducers. A full list of CYP3A inhibitors and inducers can be found here: http://www.fda.gov/drugs/developmentapprovalprocess/developmentresources/druginteractionslabeling/ucm093664.htm#4
   6. Current use or planned use of antibiotics and/or corticosteroids that may interact with levonorgestrel
   7. Non-therapeutic injection drug use in the 12 months prior to Enrollment
   8. Post-exposure prophylaxis (PEP) for HIV exposure within the 3 months prior to Enrollment
   9. Pre-exposure prophylaxis (PrEP) for HIV prevention within the 3 months prior to Enrollment
   10. Last pregnancy outcome less than 60 days prior to Enrollment
   11. Gynecologic or genital procedure (e.g., tubal ligation, dilation and curettage, piercing) 45 days or less prior to Enrollment Note: Pap test at the Screening Visit, colposcopy and cervical biopsies for evaluation of an abnormal Pap test as well as IUD insertion/removal are not exclusionary.
   12. Currently breastfeeding or planning to breastfeed during the study period
7. Any Grade 2 or higher laboratory abnormalities and any of the following Grade 1 laboratory abnormalities at the Screening Visit+:

   1. AST*
   2. ALT*
   3. Creatinine*
   4. Hemoglobin*
   5. Platelet count* Note: Otherwise eligible participants with an exclusionary laboratory result may be re-tested and may be enrolled/randomized after the findings have improved to a non-exclusionary severity grading or resolved within 90 days of providing informed consent for screening. Results of safety laboratory testing performed at the Enrollment Visit are expected to be received after the Enrollment Visit, and thus will not be exclusionary. Abnormal results will be noted as pre-existing conditions, and may result in product discontinuation, per IoR discretion as per Section 7.2.1 of the protocol.

      * DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events Corrected Version 2.1, July 2017, and/or Addendum 1 (Female Genital Grading Table for Use in Microbicide Studies [Dated November 2007])53 +This DAIDS table can be found in the SPM
8. Has any other condition that, in the opinion of the IoR/designee, would preclude informed consent, make study participation unsafe, complicate the interpretation of study outcome data, or otherwise interfere with achieving the study objectives including any significant uncontrolled active or chronic medical condition.
9. Be a site staff member with delegated study responsibilities or a family member of, or have a close relationship with, a site staff member with delegated study responsibilities.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2024-10-07 (Actual); Study Completion 2024-10-07 (Actual)

PRIMARY OUTCOMES:
Evaluate pharmacokinetics by assessing changes in baseline of DPV and LNG concentrations in plasma | 90 days (3 cycles, one cycle is approximately 30 days of continuous use)
  DPV and LNG concentrations in plasma
Evaluate pharmacokinetics by assessing changes in baseline of DPV and LNG concentrations in cervicovaginal fluid | 90 days (3 cycles, one cycle is approximately 30 days of continuous use)
  DPV and LNG concentrations in cervicovaginal fluid

SECONDARY OUTCOMES:
The safety of two DPV-LNG vaginal ring formulations | 90 days
  Incidence of Grade 2, grade 3 or higher genitourinary adverse events as defined by the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected v2.1 July 2017, or Addendum 1 Female Genital Grading Table for Use in Microbicide Studies
Assessing vaginal bleeding patterns associated with the two DPV-LNG vaginal ring formulations | 90 days
  Total number of days bleeding/spotting by participant self-report in a diary card
Assessing vaginal bleeding patterns associated with the two DPV-LNG vaginal ring formulations | 90 days
  Total number of bleeding/spotting episodes by participant self-report in a diary card
Frequency of study vaginal ring removal (voluntary and involuntary) | 90 days (3 cycles, one cycle is approximately 30 days of continuous use)
  Self-reported attitudes about ring attributes, use regimens and tolerability by completing an acceptability questionnaire. Residual drug levels (DPV and LNG) in returned vaginal rings
Duration of study vaginal ring removal | 90 days (3 cycles, one cycle is approximately 30 days of continuous use)
  Self-reported attitudes about ring attributes, use regimens and tolerability by completing an acceptability questionnaire. Residual drug levels (DPV and LNG) in returned vaginal rings

CONTACTS AND LOCATIONS:
Overall Officials: John Steytler, MBChB, Study Chair — IPM SA NPC
Locations (2):
- United States (2):
  - Oregon Health & Science University, Portland, Oregon
  - UPMC Magee-Womens Hospital, Center for Family Planning Research, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No